CLINICAL TRIAL: NCT02431130
Title: Low-fidelity Simulation to Teach Anesthetists' Non-technical Skills in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Patricia Livingston, Medical Director, Global Health Office of Anesthesia, Dalhousie University
Other Study IDs: 2011-2596
Record Dates: First submitted 2015-04-23; First posted 2015-04-30 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Training Program

ARMS (2):
- Low-fidelty instructor driven simulation training (Experimental): participants receive simulation training
  Interventions: Other: low-fidelity instructor driven simulation training
- No simulation training (No Intervention)

INTERVENTIONS:
Other: low-fidelity instructor driven simulation training
  Arms: Low-fidelty instructor driven simulation training

SUMMARY:
The goal of this study is to examine whether low-fidelity instructor-driven simulation can provide effective teaching of anesthetists' non-technical skills in a developing world context. Human factors, such as communication, planning, and team working are considered nontechnical skills which contribute greatly to patient safety in "complex hazardous systems" such as aviation, nuclear power industry, and operating rooms. Simulation began in the aviation industry to train pilots in human factors. In the past two decades simulation has been valued in medical education as it allows the learner to rehearse skills in an environment that is similar to the workplace but without the threat of harm to patients. High Fidelity simulators involve computer driven interactive mannequins that recreate an authentic environment. This has been used successfully to teach anesthetists' non-technical skills (ANTS) such as: decision making, team working, task management, and situation awareness. Anesthetists' non-technical skills are particularly important in developing countries where the shortage of supplies, equipment, and qualified personnel can lead to a perilous working environment making team work and communication vital for patient safety. The costs of high fidelity simulation are prohibitive for many developing countries. This study seeks to examine whether low fidelity instructor driven simulation can provide an effective intervention to teach anesthetists' non-technical skills in Rwanda. If found to be effective, this method of training could be applied to other developing countries to improve non-technical skills for anesthesia providers with the goal of making surgery safer.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia providers (resident or technician) that provides anesthesia for caesarean section

Exclusion Criteria:

* anesthesia providers that do not provide anesthesia for caesarean section

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Improvement in overall ANTS score after simulation training | two weeks after training